CLINICAL TRIAL: NCT01275664
Title: Pilot Study of Standard Therapy for Prevention of Nausea and Emesis Associated With First Line Post-Operative Intraperitoneal Chemotherapy
Brief Title: Granisetron, Aprepitant, and Dexamethasone in Preventing Nausea and Vomiting in Patients Receiving Chemotherapy for Stage II, III, or IV Ovarian Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to no patient population available
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GOG-0272; NCI-2011-02660 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000692516; GOG-0272 (Other: NRG Oncology); GOG-0272 (Other: DCP); GOG-0272 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Results first posted 2018-04-12 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2017-05

CONDITIONS: Nausea and Vomiting; Ovarian Brenner Tumor; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Cystadenocarcinoma; Stage II Ovarian Cancer; Stage IIA Fallopian Tube Cancer; Stage IIA Ovarian Cancer; Stage IIB Fallopian Tube Cancer; Stage IIB Ovarian Cancer; Stage IIC Fallopian Tube Cancer; Stage IIC Ovarian Cancer; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Primary Peritoneal Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Primary Peritoneal Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Nausea; Vomiting; Brenner Tumor; Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Chemotherapy, Adjuvant; Aprepitant; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Granisetron

ARMS (1):
- Treatment (granisetron, dexamethasone, aprepitant) (Experimental): Patients apply one patch of granisetron transdermal system to the upper outer arm on day 0 (at least 24 hours before intraperitoneal [IP] platinum therapy). Patients then receive dexamethasone PO on days 1-4, aprepitant IV over 15 minutes on day 1 (30 minutes before IP platinum therapy), and aprepitant PO on days 2-3.
  Interventions: Procedure: Adjuvant Therapy; Drug: Aprepitant; Drug: Carboplatin; Drug: Cisplatin; Drug: Dexamethasone; Drug: Granisetron Transdermal Patch; Procedure: Management of Therapy Complications; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Adjuvant Therapy — Ancillary studies
  Other Names: adjunct therapy; adjunctive therapy
Drug: Aprepitant — Given IV and PO
  Other Names: Emend; L-754030; MK-0869; ONO-7436
Drug: Carboplatin — Given IP
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IP
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Granisetron Transdermal Patch — Apply one patch to upper arm
  Other Names: Granisetron Transdermal System; Sancuso
Procedure: Management of Therapy Complications — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial is studying how well granisetron, aprepitant, and dexamethasone work in preventing nausea and vomiting in patients receiving chemotherapy for stage II, stage III, or stage IV ovarian cancer. Granisetron patch, aprepitant and dexamethasone may help lessen or prevent nausea and vomiting in patients receiving chemotherapy for stage II, stage III, or stage IV ovarian cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the frequency of chemotherapy-induced nausea and vomiting based on complete response (no vomiting and no use of rescue therapy) during the 6 days following intraperitoneal (IP) chemotherapy for the 3-day regimen of aprepitant (both injection and capsules) in combination with granisetron transdermal system and dexamethasone in ovarian cancer patients receiving IP cisplatin OR IP carboplatin.

SECONDARY OBJECTIVES:

I. To evaluate possible endpoints for the chemotherapy-induced nausea and vomiting, including:

* Functional Living Index-Emesis (FLIE) questionnaire scores
* Mean vomiting, nausea and total FLIE scores and changes from baseline in FLIE scores
* Percentages of patients with no impact on daily living (NIDL), i.e. > 108/126 total FLIE score II. To describe the timing of nausea and vomiting that may guide modifications to the standard regimen.

OUTLINE: This is a multicenter study.

Patients apply one patch of granisetron transdermal system to the upper outer arm on day 0 (at least 24 hours before intraperitoneal [IP] platinum therapy). Patients then receive dexamethasone orally (PO) on days 1-4, aprepitant IV over 15 minutes on day 1 (30 minutes before IP platinum therapy), and aprepitant PO on days 2-3.

Patients complete the Functional Living Index--Emesis (FLIE) and a symptom diary at baseline and on days 3 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ovarian epithelial, fallopian tube, or primary peritoneal carcinoma

  * Stage II, III, or IV disease with optimal (=< 1 cm residual disease) or suboptimal residual disease
  * All patients must have a procedure for determining diagnosis of epithelial ovarian, fallopian tube, primary peritoneal, with appropriate tissue for histologic evaluation
  * The minimum surgery required is an abdominal surgery providing tissue for histologic evaluation and establishing and documenting the primary site and stage, as well as a maximal effort at tumor debulking; if additional surgery was performed, it should have been in accordance with appropriate surgery for ovarian or peritoneal carcinoma described in the Gynecologic Oncology Group (GOG) Surgical Procedures Manual
* Patients with the following histologic epithelial cell types are eligible:

  * Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified (N.O.S.)
  * However, the histologic features of the tumor must be compatible with a primary Müllerian epithelial adenocarcinoma; if doubt exists, it is recommended that the investigator should have the slides reviewed by an independent pathologist prior to entry
  * Patients may have co-existing endometrial cancer so long as the primary origin of invasive tumor is ovarian or peritoneal for clarification of synchronous primary endometrial cancer
* Patients receiving the initial course of chemotherapy including

  * Paclitaxel 135 mg/M2 IV over 3 hours on day 1 and
  * Cisplatin 75 mg/M2 IP on day 2 OR
  * Paclitaxel 80 mg/m2 IV days 1, 8 and 15 and
  * Carboplatin AUC 6 IP on day 1
* Prothrombin time (PT) such that international normalized ratio (INR) is < 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin)
* Partial thromboplastin time (PTT) < 1.5 times the upper limit of normal (heparin, lovenox or alternative anticoagulants are acceptable)
* Patients with a GOG Performance Status of 0, 1, or 2
* Patients who are able to read, understand and write English; if FLIE which has been translated into other languages, and validated, becomes available, then patients speaking these languages can be enrolled if translation of the symptom diary can be arranged dependent on availability of suitable translators
* Patients who are able to complete the assessments
* Patients who are able to comply with the anti-emetic therapy
* Patients must have met pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients who are known to be hypersensitive to aprepitant, granisetron or any of the components of the patch or to dexamethasone
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor including neo-adjuvant chemotherapy for their ovarian or primary peritoneal cancer are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients who are pregnant or nursing; to date, no fetal studies in animals or humans have been performed; the possibility of harm to a fetus is likely
* Patients with clinical symptoms or signs of gastrointestinal obstruction and/ or those who require parenteral hydration and/or nutrition; patients with history or current diagnosis of inflammatory bowel disease are not eligible
* Patients with medical history or conditions not otherwise previously specified which in the opinion of the investigator should exclude participation in this study; examples of this would be hearing loss or neuropathy which would prevent tolerance to cisplatin, and paclitaxel administration; the investigator should feel free to consult the Study Chair or Study Co-Chairs for uncertainty in this regard
* Patients who, in the opinion of the treating physician, have a medical condition, or currently take medications, which are felt to contraindicate safe or effective administration of the standard three drug anti-emetic regimen used in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-06; Primary Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Plaxe, Principal Investigator — NRG Oncology
Locations (2):
- United States (2):
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Women and Infants Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was opened to patient entry on June 13, 2011 and was closed to accrual on December 12, 2011. The trial closed early because enrollment into this study was dependent on accruing patients simultaneously with GOG 252 (NCT00951496). When GOG 252 closed, there was no patient population to recruit from for this study.
Period: Overall Study
Arm/Group | Treatment (Granisetron, Dexamethasone, Aprepitant)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Treatment (Granisetron, Dexamethasone, Aprepitant)
Number analyzed (Participants) | 4
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 0
  50-59 years | 1
  60-69 years | 2
  70-79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Control Defined as no Vomiting and no Use of Rescue Medications (for Nausea or Emesis)
Description: Number of participants who had complete control defined by no vomiting
Time Frame: During the 6 days following chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Granisetron, Dexamethasone, Aprepitant)
Number analyzed (Participants) | 4
Participants | 1

2. Secondary Outcome: Change in Vomiting, Nausea and Total FLIE Scores
Time Frame: Baseline to day 6
Population: Data was not collected. Funding withdrawn.
Arm/Group | Treatment (Granisetron, Dexamethasone, Aprepitant)
Number analyzed (Participants) | 0

3. Secondary Outcome: Frequency of Adverse Effects as Assessed by the NCI CTCAE v 4.0
Description: Adverse events at least possibly related to treatment
Time Frame: Up to day 6
Population: All eligible and evaluable subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Granisetron, Dexamethasone, Aprepitant)
Number analyzed (Participants) | 4
Participants
  Constipation | 1
  Fatigue | 1
  Diarrhea | 1
  Hyponatremia | 1
  Alanine Aminotransferase Increased | 1
  GGT Increased | 1

4. Secondary Outcome: Mean and Standard Deviation of Vomiting, Nausea, and Total FLIE Scores
Time Frame: Baseline
Population: Data not collected. Funding withdrawn
Arm/Group | Treatment (Granisetron, Dexamethasone, Aprepitant)
Number analyzed (Participants) | 0

5. Secondary Outcome: Percentages of Patients With NIDL Based on FLIE
Time Frame: Up to day 6
Population: Data not collected. Funding withdrawn.
Arm/Group | Treatment (Granisetron, Dexamethasone, Aprepitant)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Assessed day 6 while on treatment and up to 30 days after day 6.
Arm/Group | Treatment (Granisetron, Dexamethasone, Aprepitant)
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Granisetron, Dexamethasone, Aprepitant) (N=4)
Anemia (Blood and lymphatic system disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Mucositis Oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Platelet Count Decreased (Investigations) | 1
Ggt Increased (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 2
White Blood Cell Decreased (Investigations) | 2
Aspartate Aminotransferase Increased (Investigations) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less